CLINICAL TRIAL: NCT04208100
Title: Pilot Evaluation of the Lutronic PicoPlus System for the Treatment of Benign Pigmented Lesions of the Hands
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CynosureLutronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: L18007
Record Dates: First submitted 2019-12-17; First posted 2019-12-23 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Benign Pigmented Lesions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: PicoPlus — The PICOPLUS Laser System (K173700) is indicated for use in surgical and aesthetic applications in the medical specialties of dermatology and general and plastic surgery. The 595nm and 660nm wavelengths of the Lutronic PicoPlus Laser system are used for the treatment of benign pigmented lesions.

SUMMARY:
Prospective, multi-site, non-randomized study of up to 40 treated subjects; subjects enrolled may be greater than subjects treated.

DETAILED DESCRIPTION:
Subjects will be enrolled to ensure a minimum number of subjects by skin type participate in the study as follows: FST I-II, at least 5 subjects; FST III, at least 10 subjects; FST IV, at least 5 subjects. Additionally, up to 20 training subjects will be enrolled that will be excluded from efficacy analysis, but will be included in safety analysis.

Standardized baseline and follow-up images will be taken using the sites' preferred camera system. No pre-treatment medication prior to study treatment.

Phase I: Study subjects will receive up to three treatments with the PicoPlus with the 595nm on one hand and the 660nm on the other hand. Subjects will receive the same wavelength for all treatments on each specific hand; treatments will alternate by subjects between the left side getting treated with the 595nm and the right side getting treated with the 660nm depending on enrollment. Treatments will be 30+7 days apart up to three treatments until desired clearance has been achieved.

Phase II: Up to 2 balancing treatments may be done if needed based on the investigator's discretion to achieve equal clearance on each hand utilizing the wavelength of the investigator's choice. Phase II will not be considered for efficacy endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 years and older.
2. Subject in good health.
3. Fitzpatrick Skin Type I to IV.
4. Presence of benign pigmented lesions on hands.
5. Understands and accepts the obligation not to undergo any other procedures in the treatment area.
6. Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
7. Subjects of childbearing potential must have a negative urine pregnancy test result and must not be lactating at the Screening Visit and be willing and able to use an acceptable method of birth control (e.g. barrier methods used with a spermicidal agent, hormonal methods, IUD, surgical sterilization, abstinence) during the study. Women will not be considered of childbearing potential if one of the following conditions is documented on the medical history:

   1. Postmenopausal for at least 12 months prior to study;
   2. Without a uterus and/or both ovaries; or
   3. Bilateral tubal ligation at least six months prior to study enrollment.
8. Absence of physical or psychological conditions unacceptable to the investigator.
9. Willingness and ability to provide written informed consent and HIPAA authorization prior to performance of any study-related procedure.

Exclusion Criteria:

1. Healing disorders such as those caused by diabetes mellitus, connective tissue disease, radiation therapy, or chemotherapy.
2. Subjects with a history of photosensitivity or diseases which may be stimulated by light at the wavelengths used, such as history of systemic Lupus Erythematosus, Pophyia, and Epilepsy.
3. History of chronic drug or alcohol abuse.
4. Inability to understand the protocol or to give informed consent.
5. Subjects with a history of skin cancer or current condition of any other type of cancer or pre-malignant moles.
6. Subjects who are pregnant, nursing, or anticipate a pregnancy during the length of the trial.
7. History of keloid formation.
8. Subjects with tattoos on the backs of the hands in the treatment area.
9. History of surgical or cosmetic treatments in exposure area within the past six months.
10. History of tanning or use of self-tanners in the past 4 weeks.
11. History of treatments that may irritate the skin in the treatment area such as depilatories, harsh chemicals, etc.) in the past 2 weeks.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Pigmentary Clearance | 30 days
  Percentage of pigmentary clearance by each wavelength in standard photographs from the 30-day visit post the last treatment in Phase I of the study using a score of 0-4, representing poor 0-24%, fair 25-49%, good 50-74%, excellent 75-95%, and complete 95%+ improvement was given at the day 30 follow-up visit post the last treatment as determined by three blinded physician evaluators comparing the baseline vs 30-day follow-up visit photographs.

SECONDARY OUTCOMES:
Clinician Global Aesthetic Scale | 30 days
  The Principal Investigator, sub-investigator or qualified clinician delegated by the principal investigator, will complete a Clinician Global Aesthetic Improvement Scale assessing overall aesthetic improvement by wavelength at the 30-day visit following the last treatment visit for Phase I of the study. Scale ranging 1-Very Much Improved and 5-Worse.
Subject Global Aesthetic Scale | 30 days
  2. The subject will complete a SGAIS assessing overall aesthetic improvement by wavelength at the 30-day visit following the last treatment visit for Phase I of the study. Scale Ranging 1-Very Much Improved and 5-Worse.

OTHER OUTCOMES:
Patient Satisfaction Questionnaire | 30 days
  The subject will complete a Patient Satisfaction Questionnaire by wavelength at the 30-day visit following the last treatment visit for Phase I of the study. There are 4 questions.
Pain Scale | 30 days
  During all study treatments, the subject's pain levels will be monitored using a validated Numeric Rating Scale ranging from 0-10. The maximum and average pain score will be recorded by wavelength.

CONTACTS AND LOCATIONS:
Locations (1):
- William LoVerme, MD, Billerica, Massachusetts, United States